CLINICAL TRIAL: NCT06869707
Title: Multidisciplinary Approach to Nutritional Support for Oncological Patients - NUTRACARE PROJECT
Acronym: NUTRACARE
Status: Active, not recruiting | Type: Observational
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Sponsor
Other Study IDs: 4982
Record Dates: First submitted 2025-03-06; First posted 2025-03-11 (Actual); Last update posted 2025-03-11 (Actual); Status verified 2025-03

CONDITIONS: Gastrointestinal Neoplasms
MeSH Terms: conditions — Gastrointestinal Neoplasms

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Malnutrition correlated to increased perioperative morbidity occurs in patients with gastrointestinal malignancies.

Adherence guidelines for nutritional assessment and support in oncological patients is unfortunately very low.

The aim of the study is to improve clinical practice by using and testing the digital platform NUTRACARE in 5 different Centers.

DETAILED DESCRIPTION:
After being informed about the study, all the patients undergoing elective surgery or first cycle of neoadjuvant or adjuvant therapy giving written informed consent will be screened by the surgeon or the oncologist and the NRS-2002 (Nutrition Risk Screening) will be administered.

Patients who will be assessed at risk will be notified to the center nutritionist.

ELIGIBILITY:
Inclusion Criteria:

* <18 years
* ECOG grade 0-2
* Patients undergoing elective surgery or first cycle of chemotherapy (neoadjuvant or adjuvant) for staged I-III colorectal, hepatobiliary-pancreatic and oesophago-gastric cancers

Exclusion Criteria:

* >18 years
* Pregnancy
* Emergency
* ECOG ≥ 3
* M+
* Peritoneal involvement
* Inability to provide informed consent
* Informed consent refusal

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with gastrointestinal neoplasms
Sampling Method: Non-Probability Sample
Enrollment: 85 (Actual)
Dates: Start 2023-07-03 (Actual); Primary Completion 2023-07-17 (Actual); Study Completion 2025-07-01 (Estimated)

PRIMARY OUTCOMES:
Nutritional intervention | 15 days
  Number and type of nutritional interventions required

SECONDARY OUTCOMES:
Complications | up tp 30 days
  Number and severity of surgical and oncological complications

CONTACTS AND LOCATIONS:
Overall Officials: Domenico D'Ugo, Principal Investigator — Fondazione Policlinico Universitario A. Gemelli, IRCCS
Locations (1):
- Fondazione Policlinico Universitario A. Gemelli, IRCCS, Roma, Italy